CLINICAL TRIAL: NCT02541617
Title: Hub and Spoke, Comparative Outcomes for Parkinson's Disease Treated With Deep Brain Stimulation
Acronym: Hub&Spoke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Vanderbilt University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Fenna Phibbs, Assistant Professor of Neurology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150174
Record Dates: First submitted 2015-04-22; First posted 2015-09-04 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2016-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Movement Disorder Center (Active Comparator): Device programming, Deep Brain stimulator will be programmed at the implanting center, standard of care
  Interventions: Procedure: Standard of care
- Programming by community Neurologist (Experimental): Device programming, Deep Brain Stimulator will be programmed by community Neurologist
  Interventions: Procedure: Programming by community Neurologist

INTERVENTIONS:
Procedure: Programming by community Neurologist — Deep Brain stimulator with be programmed by a community Neurologist
  Arms: Programming by community Neurologist
Procedure: Standard of care — Deep Brain Stimulator will be programmed with at the implanting movement disorders center
  Arms: Movement Disorder Center

SUMMARY:
Outcomes study to test the hypothesis that patients first identified by community-based neurologists, implanted by a networked movement disorders center, and then managed by the same community-based neurologist will have clinical outcomes comparable to movement disorders centers.

DETAILED DESCRIPTION:
The proposed outcomes study is a prospective, randomized, multicenter, single blind, non-inferiority clinical trial comparing the safety and efficacy of deep brain stimulation therapy applied in a community-based model for 62 subjects with Parkinson's disease appropriate for STN DBS therapy.

Eight community-based private neurology practices will be networked to Vanderbilt University Medical Center (VUMC). Neurologists for each practice will attend structured educational programs offered by Medtronic in the identification, selection, and management of Parkinson's disease patients with DBS therapy. Following this educational program, each practice will identify subjects for implantation VUMC. Following screening and baseline visits at VUMC, appropriate patients will be implanted with bilateral subthalamic nucleus deep brain stimulating therapy. The initial post-operative programming will be done at VUMC four weeks after implantation. 8 subjects will then be equally randomized with half being followed for long-term management by the community-based neurologist. The other half will be followed at VUMC.

All subsequent outpatient evaluation management of medications and deep brain stimulation will be managed per standard of care at the location assigned by randomization, community-based private neurology practice or VUMC.

All subjects will be enrolled during the first 24 months of the study. Follow-up evaluations at 12 months will be performed at VUMC. Each patient identified by the community-based neurologist for implantation will be assessed at VUMC. This assessment will include a videotaped off and on UPDRS III rating, neuropsychological testing, and appropriateness as outlined in the patient selection educational program. Patients will be implanted by bilateral subthalamic nucleus deep brain stimulation therapy within 120 days of their initial assessment. The initial post-operative programming will be performed four weeks post-operatively, this is all standard of care.

Subjects will then be randomized to be either managed by their community-based neurologist or at VUMC. Follow-up evaluations at 12 months will include a videotaped on and off UPDRS rating and neuropsychological testing, anti-parkinson medication dosages, and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a clinical diagnosis of probable idiopathic PD. The diagnosis will be based upon the presence of at least three of four clinical features according to diagnostic utility (Resting Tremor, Bradykinesia, Rigidity, Asymmetric Onset) and an absence of clinical features suggestive of an alternative diagnosis.
2. Demonstrated response to dopaminergic therapy. In order to exclude patients with a possible alternative diagnosis, all subjects included in the study must have demonstrated a good response to DA drugs, defined as demonstrating at least 30% improvement in parkinsonian motor signs, based upon the UPDRS motor examination subscore, following the administration of their DA drug(s) during the screening neurological examination.
3. Advanced Parkinson's disease.
4. No contraindications to surgery.
5. Age between 50 and 75 years old.
6. Available for follow-up for the entire duration of the study.
7. Informed Consent: The subject understands the risks, benefits, and alternatives to the study procedures and participation in the study.
8. MRI within normal range for age

Exclusion Criteria:

1. Evidence of an alternative diagnosis or secondary parkinsonism, as suggested by features unusual early in the clinical course: Prominent postural instability, freezing phenomena, or hallucinations unrelated to medications in the first 3 years after symptom onset; dementia preceding motor symptoms; supranuclear gaze palsy (other than restriction of upward gaze) or slowing of vertical saccades in the first year; severe, symptomatic dysautonomia unrelated to medications; documentation of a condition known to produce parkinsonism and plausibly connected to the subject's symptoms (such as suitably located focal brain lesions or neuroleptic use within the past 6 months)
2. Uncontrolled medical condition or clinically significant medical disease that would increase the risk of developing pre- or postoperative complications (e.g., significant cardiac or pulmonary disease, uncontrolled hypertension).
3. Evidence of dementia
4. Major psychiatric disorder
5. Previous brain operation or injury.
6. Active participation in another clinical trial for the treatment of PD.
7. Patients who have demand cardiac pacemakers or who have medical conditions that require repeat MRI scans.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
UPDRS part IV | one year
  Change in score from baseline, complication of medical therapy for Parkinson's disease

SECONDARY OUTCOMES:
UPDRS | One Year
  Change from baseline, composite score of all 4 parts of the UPDRS
PDQ-39 | One year
  Change from baseline in quality of life
Obeso Dyskinesia Rating Scale | One year
  Change from baseline, involuntary movements caused by Parkinson's disease treatment
Hoehn and Yahr rating | One year
  Change from baseline, in stage of disease
Schwab and England ADL score | One year
  Change from baseline, signs and symptoms of depression
Parkinson's medication in LEDD | One year
  Change from baseline in total Parkinson's disease medications
DBS voltage/current | One year
  One year settings of DBS system
DBS electrode configuration | One year
  One year settings of DBS system
DBS pulse width | one year
  One year settings of DBS system
DBS frequency | one year
  One year settings of DBS system

CONTACTS AND LOCATIONS:
Overall Officials: Fenna T Phibbs, MD, Principal Investigator — Vanderbilt Univeristy Medical center